CLINICAL TRIAL: NCT02532946
Title: Bedsider.Org in Post-abortion Contraceptive Counseling: A Mixed Methods Study
Acronym: Bedsider
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-31382
Record Dates: First submitted 2015-03-09; First posted 2015-08-26 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bedsider counseling group (Experimental): Women exposed to: Bedsider.org counseling will be offered a computer or tablet at check-in to clinic. The outcome measure is measured at the patient's surgical abortion procedure appointment, or at medical abortion follow-up, which can range up to 10 days after enrollment
  Interventions: Behavioral: Bedsider.org counseling
- Routine counseling group (No Intervention): Women were given counseling in the providers' usual practice style. They were given a card with Bedsider.org's web address along with the counseling.

INTERVENTIONS:
Behavioral: Bedsider.org counseling — Contraceptive counseling was done while women kept the computer/tablet throughout their visit to facilitate discussion of website information with their providers.
  Arms: Bedsider counseling group

SUMMARY:
This is a mixed methods study, incorporating a randomized controlled trial and a qualitative provider focus group, to evaluate contraceptive counseling aided by www.Bedsider.org in patients seeking first-trimester abortion. The primary outcome is the uptake of long-acting reversible contraception in women seeking induced abortion.

DETAILED DESCRIPTION:
Nearly half of pregnancies among American women are unintended, and about 4 in 10 of these are terminated by abortion. Unmet need for family planning is the cause for induced abortion, and those women seeking induced abortion are a high risk for repeat abortion. Family planning services are of paramount importance to this population, and evidence shows that high-quality family planning counseling and provision of methods prior to discharge from a care facility improve uptake and continuation of methods. In a recent study, oral contraceptive pills, a transdermal patch, or a vaginal ring had a risk of contraceptive failure that was 20 times as high as the risk among those using long-acting reversible contraception (IUD or implant).

We plan to randomize preoperative clinic days to either provider counseling aided by Bedsider.org or routine provider counseling, and compare the types of contraceptive methods that are chosen in each group, with the primary outcome being uptake of long-acting reversible contraception (intrauterine device or implant). The secondary outcome is satisfaction with contraceptive counseling in both groups.

We also plan to conduct a qualitative focus group study of provider perspectives of this counseling tool after completion of the randomized trial. Materials related to the qualitative portion of the study will be submitted in a separate amendment. No Follow-up is needed.

EXPECTED OUTCOMES AND DISSEMINATION OF FINDINGS The goal of the study is to assess the feasibility and effectiveness of using a web-based contraception tool in a unique family planning clinic serving high-risk patients with expert family planning providers. After assessing feasibility, utility, and effectiveness in our practice setting, we hope to spread the use of bedsider.org to the entirety of the outpatient clinic, which includes general obstetrics and gynecology patients and providers.

After completion of the study, we plan to submit our findings for presentation at a national meeting, and submit a manuscript for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Seeking medical or surgical pregnancy termination
* 12 weeks gestation or less

Exclusion Criteria:

* Early pregnancy failure
* Medical contraindications to any contraceptive methods as based on CDC Medical Eligibility Criteria

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 346 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Uptake, as measured by questionnaire, of long-acting reversible contraception (LARC) in 18-29 women seeking induced abortion | Up to 10 days
  Decision on contraceptive tool selected: LARC - Yes or No

SECONDARY OUTCOMES:
Satisfaction with a web based tool as measured by a Likert scale | Up to 10 days
  Short Questionnaire with likeret scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Soanlkar, MD MPH, Principal Investigator — Hospital of the University of Pennsylvania Department of Obstetrics and Gynecology

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed journal

REFERENCES:
- See also: Bedsider site — https://bedsider.org/